CLINICAL TRIAL: NCT04221217
Title: Phase 3 Long-term Study to Evaluate the Safety and Efficacy of MND-2119 in Patients With Hypertriglyceridemia
Brief Title: Long-term Safety and Efficacy Study of MND-2119 in Patients With Hypertriglyceridemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MND2119H41; JapicCTI (Registry Identifier: JapicCTI-205100)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2020-09

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MND-2119 2g (Experimental): MND-2119 2 g, orally, once daily after breakfast for 52 weeks.
  Interventions: Drug: Icosapent
- MND-2119 4g (Experimental): MND-2119 4 g, orally, once daily after breakfast for 52 weeks.
  Interventions: Drug: Icosapent

INTERVENTIONS:
Drug: Icosapent — Icosapent (MND-2119) capsules.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of MND-2119 at a dose of 2g/day or 4g/day for 52 weeks in patients with hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed with hypertriglyceridemia.
2. Participants with values of fasting triglyceride level are 150 mg/dL or higher and less than 500 mg/dL.

Exclusion Criteria:

1. Participants who have confirmed myocardial infarction and angina pectoris within 6 months.
2. Participants who have aortic aneurysm or has received aortic aneurysmectomy within 6 months.
3. Participants with, or with a history of, pancreatitis.
4. Participants who have a history or complication of a clinically significant hemorrhagic disease within 6 months.
5. Participants taking both anti-coagulants and anti-platelets.
6. Participants receiving dual antiplatelet therapy (DAPT).
7. Participants taking direct oral anticoagulants (DOAC) or warfarin.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | 52 Weeks

SECONDARY OUTCOMES:
Number of Participants With Adverse Drug Reactions (ADRs) | 52 Weeks
Actual Value and Percent Change From Baseline in Triglyceride | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Actual Value and Percent Change From Baseline in Total Cholesterol | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Actual Value and Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Actual Value and Percent Change From Baseline in High-Density Lipoprotein-Cholesterol (HDL-C) | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Actual Value and Percent Change From Baseline in Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) | Baseline and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Takuya Mori, Study Director — Mochida Pharmaceutical Company, Ltd.
Locations (1):
- Mochida Investigational sites, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No